CLINICAL TRIAL: NCT00332436
Title: Safety and Efficacy Study of Brimonidine/Timolol Fixed Combination in Patients With Glaucoma or Ocular Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Therapeutic Area Head, Allergan, Inc
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 190342-013T
Record Dates: First submitted 2006-05-30; First posted 2006-06-01 (Estimated); Last update posted 2011-05-30 (Estimated); Status verified 2011-05

CONDITIONS: Ocular Hypertension
MeSH Terms: conditions — Ocular Hypertension | interventions — Brimonidine Tartrate

INTERVENTIONS:
Drug: brimonidine/timolol fixed combination

SUMMARY:
The purpose of this study is to assess the safety and efficacy of Brimonidine/Timolol Fixed Combination in patients with glaucoma or ocular hypertension

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of ocular hypertension or chronic glaucoma in both eyes
* Patient requires IOP-lowering drug in both eyes

Exclusion Criteria:

* Uncontrolled medical condition
* Contraindication to beta-adrenoceptor antagonist or brimonidine therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 586 (Actual)
Dates: Start 1999-12; Primary Completion 2001-11 (Actual); Study Completion 2001-11 (Actual)

PRIMARY OUTCOMES:
IOP

CONTACTS AND LOCATIONS:
Locations (1):
- Louisville, Kentucky, United States